CLINICAL TRIAL: NCT06824090
Title: Investigation of Tonus, Stiffness and Elasticity of Hand and Wrist Muscles in Intensive Smartphone Use
Brief Title: Tonus, Stiffness and Elasticity of Hand and Wrist Muscles in Smartphone Addiction
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hazel Çelik Güzel, Assist. Prof. Dr, Bandırma Onyedi Eylül University
Other Study IDs: 2024-114
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Muscle Biomechanics; Smartphone Addisction
Keywords: smartphone; tonus; stiffness; elasticity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Smartphone Addiction Scale-Short Form — Smartphone Addiction Scale-Short Form: In our study, the Smartphone Addiction Scale-Short Form will be filled out in order to evaluate the intensity of smartphone use of students, and the daily duration of smartphone use will be recorded. The scale is a 6-point Likert-type scale consisting of 10 items used to measure the risk of smartphone addiction. Scores obtained from the scale vary between 10-60 and an increase in the score indicates an increased risk for smartphone addiction. The cut-off score of the scale was determined as 31 for men and 33 for women. In the Turkish validity and reliability study, Cronbach's alpha coefficient was found to be 0.86.
Other: Hand Grip Strength Assessment — Hand grip strength was measured with 'Saehan Hydraulic Hand Dynamometer'. Participants were informed about the correct holding position and use of the instrument. In the measured arm, the position of 90̊ flexion from the elbow joint and completely adjacent to the body was used. The participant's hand was placed in the second grip position of the dynamometer and asked to make the strongest grip he/she could make, right and left measurements were taken.
Other: Finger Lateral Grip Strength Assessment — Finger lateral grip strength was measured with 'Saehan Hydraulic pinch gauge'. Participants were informed about the correct holding position and use of the instrument. While the participant was sitting on a chair with arms supported, the shoulder was adjacent to the trunk and neutral, the elbow joint was in 90 ̊ flexion, the forearm was neutral, the wrist was in 0-30 ̊ extension and 0-15 ̊ ulnar deviation. Right and left finger lateral grip measurements were taken.
Other: Myoton Assessment — Myoton PRO device was used to objectively evaluate the biomechanical properties of the hand and wrist muscles such as tone, stiffness and elasticity. Tenar region, flexor carpi radialis, flexor carpi ulnaris, extensor digitorum, extensor carpi radialis and extensor carpi ulnaris muscles were evaluated bilaterally. Three measurements were recorded at one second intervals and the mean value was used for analysis.

SUMMARY:
The aim of this study was to investigate the tonus, stiffness and elasticity of the hand and wrist muscles in intensive smartphone use.

DETAILED DESCRIPTION:
Consent was obtained from the students with the 'Informed Voluntary Consent Form' and the sociodemographic data of the students were recorded on the previously prepared Descriptive Data Form. The students were asked to fill out the Smartphone Addiction Scale-Short Form. Before starting the clinical evaluation, anamnesis was taken from the students and their general health status, phone usage time (minutes) and exclusion criteria were questioned. Myotone evaluations of the tenar region, flexor carpi radialis, flexor carpi ulnaris, extensor digitorum, extensor carpi radialis and extensor carpi ulnaris muscles were performed. Then, the standard grip strength of the dominant and non-dominant side hand was evaluated with Saehan hand dynamometer and the lateral grip strength of the thumb was evaluated with Saehan pinchmeter.

ELIGIBILITY:
Inclusion Criteria:

* To study at Bandirma Onyedi Eylül University
* Students between the ages of 18-30 years, whose voluntary consent was obtained and who use smartphones

Exclusion Criteria:

* Individuals with musculoskeletal system problems such as fractures of the hand, fingers and upper extremities, rheumatoid disease with evidence of systemic, specific pathological conditions
* Individuals who have undergone any surgical operation related to hand, finger and upper extremity problems
* Individuals who have received hand, finger and upper extremity related physiotherapy and rehabilitation services in less than 6 months
* Individuals with diagnosed psychiatric illness.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Study Population: University students
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Smartphone Addiction Scale-Short Form | May 1, 2024- January 1, 2025
  Smartphone Addiction Scale-Short Form: In our study, the Smartphone Addiction Scale-Short Form will be filled out in order to evaluate the intensity of smartphone use of students, and the daily duration of smartphone use will be recorded. The scale is a 6-point Likert-type scale consisting of 10 items used to measure the risk of smartphone addiction. Scores obtained from the scale vary between 10-60 and an increase in the score indicates an increased risk for smartphone addiction. The cut-off score of the scale was determined as 31 for men and 33 for women. In the Turkish validity and reliability study, Cronbach's alpha coefficient was found to be 0.86.
Hand grip strength assessment | May 1, 2024- January 1, 2025
  Hand grip strength was measured with 'Saehan Hydraulic Hand Dynamometer'. Participants were informed about the correct holding position and use of the instrument. In the measured arm, the position of 90̊ flexion from the elbow joint and completely adjacent to the body was used. The participant's hand was placed in the second grip position of the dynamometer and asked to make the strongest grip he/she could make, right and left measurements were taken.
Finger lateral grip strength assessment | May 1, 2024- January 1, 2025
  Finger lateral grip strength was measured with 'Saehan Hydraulic pinch gauge'. Participants were informed about the correct holding position and use of the instrument. While the participant was sitting on a chair with arms supported, the shoulder was adjacent to the trunk and neutral, the elbow joint was in 90 ̊ flexion, the forearm was neutral, the wrist was in 0-30 ̊ extension and 0-15 ̊ ulnar deviation. Right and left finger lateral grip measurements were taken.
Myoton assessment | May 1, 2024- January 1, 2025
  Myoton PRO device was used to objectively evaluate the biomechanical properties of the hand and wrist muscles such as tone, stiffness and elasticity. Tenar region, flexor carpi radialis, flexor carpi ulnaris, extensor digitorum, extensor carpi radialis and extensor carpi ulnaris muscles were evaluated bilaterally. Three measurements were recorded at one second intervals and the mean value was used for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Balıkesir, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided